CLINICAL TRIAL: NCT02923193
Title: Randomized Study of the Shockwave Medical Peripheral Lithoplasty® System Used in Combination With DCB Versus Standard Balloon Angioplasty Used in Combination With DCB to Treat Moderate and Severely Calcified Femoropopliteal Arteries
Brief Title: Shockwave Medical Peripheral Lithoplasty System Study for PAD (Disrupt PAD III)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP 60892
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lithoplasty System followed by DCB (Experimental): Shockwave Lithoplasty® Peripheral Lithoplasty System is a lithotripsy-enhanced, low-pressure balloon dilatation of calcified, stenotic peripheral arteries in patients who are candidates for percutaneous therapy. lithoplasty
  Interventions: Device: Shockwave Lithoplasty® Peripheral Lithoplasty System; Drug: Medtronic IN.PACT (DCB)
- Medtronic IN.PACT (DCB) (Active Comparator): Medronic IN.PACT Drug Coated Balloon (DBS) is indicated for percutaneous transluminal angioplasty (PTA) in patients with obstructive disease of peripheral arteries, including patients with in-stent restenosis (ISR) and arteriovenous (AV) access to help maintain hemodialysis access in patients with end-stage renal disease.
  Interventions: Drug: Medtronic IN.PACT (DCB)

INTERVENTIONS:
Device: Shockwave Lithoplasty® Peripheral Lithoplasty System — The Shockwave Lithoplasty® System is a proprietary lithotripsy-enhanced balloon catheter that is designed to be delivered through the peripheral arterial system of the lower extremities to the site of calcified stenosis. Activating the lithotripsy within the device will generate pulsatile mechanical energy within the target treatment site, disrupt calcium within the lesion and allow subsequent dilation of a peripheral artery stenosis using low balloon pressure. The system consists of a balloon catheter with multiple integrated lithotripsy electrodes, and a generator.
  Arms: Lithoplasty System followed by DCB
Drug: Medtronic IN.PACT (DCB) — The IN.PACT Admiral DCB is an over-the-wire (OTW) balloon catheter with a drug-coated balloon at the distal tip. The drug component, referred to as the FreePac™ drug coating, consists of the drug paclitaxel and the excipient urea. The device component physically dilates the vessel lumen by PTA, and the drug is intended to reduce the proliferative response that is associated with restenosis.
  Other Names: drug coated balloon

SUMMARY:
Shockwave Medical Inc. intends to conduct a prospective, multi-center, single blind, randomized (1:1) study of Lithoplasty treatment used in combination with DCB versus standard balloon angioplasty used in combination with DCB to treat moderate and severely calcified femoropopliteal arteries. Assuming that roughly 15% of the subjects will be lost-to-follow-up, a total of up to 400 subjects (200 per treatment arm) will be enrolled in the study at up to 60 sites in Europe, the United States and New Zealand.

In addition to the randomized study, an observational study of subjects who do not meet the inclusion/exclusion criteria for the randomized study will be conducted. The objective of the observational study is to assess the real-world acute performance of the Shockwave Medical Peripheral Lithoplasty System in the treatment of calcified, stenotic, peripheral arteries.

The observational study is a prospective, multi-center, single arm observational study for subjects who do not meet the inclusion/exclusion criteria of the randomized study.

A maximum of 1500 subjects at the same 60 sites will be enrolled in the observational study. Once enrollment in the randomized portion of the study is complete, subjects may continue to be enrolled in the observational study provided they meet OS eligibility criteria.

Results for the observational study will be reported in a separate record under NCT05881421.

DETAILED DESCRIPTION:
Shockwave Medical Inc. intends to conduct a prospective, multi-center, single blind, randomized (1:1) study of Lithoplasty treatment used in combination with DCB versus standard balloon angioplasty used in combination with DCB to treat moderate and severely calcified femoropopliteal arteries. The Shockwave Medical Peripheral Lithoplasty System is indicated for lithotripsy-enhanced, low-pressure balloon dilatation of calcified, stenotic peripheral arteries in patients who are candidates for percutaneous therapy. Up to 400 subjects at 60 sites in Europe, the United States and New Zealand.

Subjects will be followed through discharge, 30 days, and 6, 12 and 24 months. DUS assessments will be completed at 12 and 24 months. Procedural success is defined as residual stenosis ≤30% without flow-limiting dissection (≥ grade D) prior to DCB or stenting by angiographic core lab.

Subjects who do not meet the randomized study inclusion and exclusion criteria, but meet the inclusion and exclusion criteria for the observational study may be enrolled in the observational study. The objective of the observational study is to assess the real-world acute performance of the Shockwave Medical Lithoplasty System in the treatment of calcified, stenotic, peripheral arteries.The observational study is a prospective, multi-center, single arm observational study for subjects who do not meet the inclusion/exclusion criteria of the randomized study. A maximum of 1500 subjects at the same 60 sites will be enrolled in the observational study. Procedural success is defined as residual stenosis ≤30% without flow-limiting dissection (≥ grade D) prior to DCB or stenting by angiographic core lab. Enrollment in the observational study is anticipated to last approximately 22 months. Subjects in the observational study will be followed through hospital discharge. Once enrollment in the randomized portion of the study is complete, subjects may continue to be enrolled in the observational study provided they meet OS eligibility criteria. Results for the observational study will be reported in a separate record under NCT05881421.

ELIGIBILITY:
Randomized Study Arm Eligibility Criteria

General Inclusion Criteria

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
3. Age of subject is greater than or equal to 18.
4. Rutherford Clinical Category 2, 3, or 4 of the target limb.
5. Estimated life expectancy >1 year.
6. Subject is a suitable candidate for angiography and endovascular intervention in the opinion of the investigator or per hospital guideline.
7. Subject is intended to undergo treatment with Lithoplasty followed by DCB, or DCB with standard balloon pre-dilatation.

   Angiographic Inclusion Criteria
8. Target lesion that is located in a native, de novo superficial femoral artery (SFA) or popliteal artery (popliteal artery extends to and ends proximal to the ostium of the anterior tibial artery).
9. Target lesion reference vessel diameter is between 4.0mm and 7.0mm by visual estimate.
10. Target lesion is ≥70% stenosis by investigator via visual estimate.
11. Target lesion length is ≤180mm for lesions 70-99% stenosed. Target lesion can be all or part of the 180mm treated zone.
12. Chronic total occlusion, lesion length is ≤100mm of the total ≤180 mm target lesion.
13. Subject has at least one patent tibial vessel on the target leg with runoff to the foot, defined as no stenosis >50%.
14. Calcification is at least moderate defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

General Exclusion Criteria

1. Rutherford Clinical Category 0, 1, 5 and 6.
2. Subject has active infection requiring antibiotic therapy.
3. Planned target limb major amputation (above the ankle).
4. History of prior endovascular or surgical procedure on the index limb within the past 30 days or planned within 30 days of the index procedure.
5. Subject has a known coagulopathy or has bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter.
6. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
7. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
8. Subject has known allergy to urethane, nylon, or silicone.
9. Myocardial infarction within 60 days prior to enrollment.
10. History of stroke within 60 days prior to enrollment.
11. History of thrombolytic therapy within two weeks of enrollment.
12. Subject has acute or chronic renal disease defined as serum creatinine of >2.5 mg/dL or >220 umol/L, or on dialysis.
13. Subject is pregnant or nursing.
14. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
15. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
16. The use of specialty balloons, re-entry or atherectomy devices.

    Angiographic Exclusion Criteria
17. In-stent restenosis within 10mm of the target zone.
18. Lesions within 10mm of the ostium of the SFA or within 10mm of the ostium of the anterior tibial artery.
19. Evidence of aneurysm or thrombus in target vessel.
20. No calcium or mild calcium in the target lesion.
21. Target lesion within native or synthetic vessel grafts.
22. Subject has significant stenosis (>50% stenosis) or occlusion of inflow tract before target treatment zone (e.g. iliac or common femoral) not successfully treated.
23. Subject requires treatment of a peripheral lesion on the ipsilateral limb distal to target site at the time of the index procedure.
24. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

Subjects who do not meet the inclusion/exclusion criteria for the randomized study may satisfy the eligibility criteria for the observational study.

Observational Study Eligibility Criteria

Inclusion Criteria

1. Subjects intended to be treated with the Shockwave Medical Peripheral Lithoplasty® System for de-novo or restenotic lesions of the femoral, ilio-femoral, popliteal, and infra-popliteal arteries.
2. Subjects presenting with claudication or CLI by Rutherford Clinical Category 2,3,4,5, or 6 of the target limb.
3. Age of subject is > 18.
4. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate, and has signed the approved study consent form.
5. Calcification is at least moderate, defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

Exclusion Criteria

1. Subjects with any medical condition that would make him/her an inappropriate candidate for treatment with Shockwave Medical Peripheral Lithoplasty® System as per Instructions for Use (IFU) or investigator's opinion.
2. Subject is already enrolled in other investigational (interventional) studies that would interfere with study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — RoMed Klinikum Rosenheim; William A Gray, MD, Principal Investigator — Main Line Health
Locations (54):
- United States (40):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Stanford Hospital, Palo Alto, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth Northern Colorado, Loveland, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Cardiovascular Research Network @ Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Advocate Health and Hospitals Corporation, Naperville, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Steward St. Elizabeth's Medical Center, Brighton, Maine
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Ascension / St. John Providence, Southfield, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Luke's Cardiovascular Consultants, Kansas City, Missouri
  - St. Luke's East Hospital, Lee's Summit, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Mount Sinai West, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - St. John Clinic, Bartlesville, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - PinnacleHealth Harrisburg Hospital, Harrisburg, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Baptist Medical Center, Memphis, Tennessee
  - St. David's Heart and Vascular dba Austin Heart, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Gefäßsambulanz, Vienna
- Germany (11):
  - Karolinen-Hospital, Arnsberg
  - Universitäts-Herzzentrum Freiburg & Bad Krozingen, Bad Krozingen
  - Sankt Gertrauden-Krankenhaus, Berlin
  - Leiter Sektion Angiologie, Bonn
  - Medizinische Klinik II, Bruchsal
  - Klinik für Gefäßmedizin, Hamburg
  - Universitätsklinikum Leipzig AoR Leipzig, Leipzig
  - Katholisches Klinikum Mainz, Mainz
  - Evangelisches Krankenhaus Mühlheim an der Ruhr, Mülheim
  - St. Franziskus Hospital, Münster
  - RoMed Klinikum Rosenheim, Rosenheim
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagpal S, Altin SE, McGinigle K, Mangalmurti SS, Adams G, Shammas NW, Mehrle A, Soukas P, Bertolet B, Lansky AJ. Sex-specific analysis of intravascular lithotripsy for peripheral artery disease from the Disrupt PAD III observational study. J Vasc Surg. 2024 Feb;79(2):358-365. doi: 10.1016/j.jvs.2023.10.058. Epub 2023 Nov 2. PMID 37925039
- [Derived] Tepe G, Brodmann M, Werner M, Bachinsky W, Holden A, Zeller T, Mangalmurti S, Nolte-Ernsting C, Bertolet B, Scheinert D, Gray WA; Disrupt PAD III Investigators. Intravascular Lithotripsy for Peripheral Artery Calcification: 30-Day Outcomes From the Randomized Disrupt PAD III Trial. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1352-1361. doi: 10.1016/j.jcin.2021.04.010. PMID 34167675
- [Derived] Adams G, Shammas N, Mangalmurti S, Bernardo NL, Miller WE, Soukas PA, Parikh SA, Armstrong EJ, Tepe G, Lansky A, Gray WA. Intravascular Lithotripsy for Treatment of Calcified Lower Extremity Arterial Stenosis: Initial Analysis of the Disrupt PAD III Study. J Endovasc Ther. 2020 Jun;27(3):473-480. doi: 10.1177/1526602820914598. Epub 2020 Apr 3. PMID 32242768
- See also: Intravascular lithotripsy for treatment of calcified, stenotic iliac arteries: A cohort analysis from the Disrupt PAD III Study — https://pubmed.ncbi.nlm.nih.gov/32147133/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Started | 153 | 153
Completed | 121 | 121
Not Completed | 32 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB) | Total
Number analyzed (Participants) | 153 | 153 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (8.0) | 71.5 (7.7) | 71.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 33 | 80
  Male | 106 | 120 | 226
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 143 | 133 | 276
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 9 | 7 | 16
  Austria | 25 | 24 | 49
  United States | 80 | 88 | 168
  Germany | 39 | 34 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural Success
Description: Procedural success is defined as residual stenosis ≤30% without flow-limiting dissection (≥ grade D) prior to DCB or stenting by angiographic core lab.
Time Frame: Peri-Procedural, approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 146 | 133
Participants | 96 | 67

2. Secondary Outcome: Number of Participants With Major Adverse Events (MAEs)
Description: * Need for emergency surgical revascularization of target limb
  * Unplanned target limb major amputation (above the ankle)
  * Symptomatic thrombus or distal emboli that require surgical, mechanical or pharmacologic means to improve flow and extend hospitalization
  * Perforations that require an intervention, including bail-out stenting
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 152 | 153
Participants | 0 | 2

3. Secondary Outcome: Clinical Success ABI
Description: Defined as ankle-brachial index ABI reported at 30 days as change from baseline. The ABI is the ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery. Ideally, this ratio should be 1.0, but is often less in a subject with peripheral arterial disease.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 140 | 135
index | .23 (.21) | .22 (.23)

4. Secondary Outcome: Clinical Success Quality of Life
Description: Defined by Quality of Life assessed by EQ5D questionnaire reported at 30 days as change from baseline. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The overall summary index (from Shaw et. al.) computed from the 5-dimension sub-scores was applied. It ranges from 0.000 to 1.000; higher scores indicate better patient-reported health status."
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 143 | 146
units on a scale | .103 (.202) | .116 (.184)

5. Secondary Outcome: Clinical Success Rutherford Category
Description: Defined as Rutherford Category reported at 30 days as change from baseline. Clinical scale identifying three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss. 0 is asymptomatic and 6 is ulcers/gangrene.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 145 | 148
units on a scale | -2.20 (1.08) | -2.27 (.99)

6. Secondary Outcome: Number of Participants With Clinically-driven Target Lesion Revascularization (TLR)
Description: Any revascularization (endovascular or surgical) within the target femoropopliteal vessel due to symptoms or drop of ABI >20% or >0.15 when compared to the 30-day ABI and associated with an angiographic lesion >50% at the target lesion site
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 152 | 153
Participants | 0 | 1

7. Secondary Outcome: Number of Participants With Major Adverse Events (MAEs)
Description: as for outcome 2
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 147 | 147
Participants | 0 | 2

8. Secondary Outcome: Clinical Success Rutherford Category
Description: Defined as Rutherford Category reported at 6 months as change from baseline. Clinical scale identifying three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss. 0 is asymptomatic and 6 is ulcers/gangrene.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 138 | 140
units on a scale | -2.35 (.91) | -2.29 (1.0)

9. Secondary Outcome: Number of Participants With Clinically-driven Target Lesion Revascularization (TLR)
Description: as for outcome 6
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 147 | 148
Participants | 4 | 1

10. Secondary Outcome: Clinical Success ABI
Description: Defined as ankle-brachial index ABI reported at 6 months as change from baseline. The ABI is the ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery. Ideally, this ratio should be 1.0, but is often less in a subject with peripheral arterial disease.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 133 | 133
units on a scale | .23 (.21) | .22 (.26)

11. Secondary Outcome: Clinical Success Quality of Life
Description: Defined by Quality of Life assessed by EQ5D questionnaire reported at 6 months as change from baseline. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The overall summary index (from Shaw et. al.) computed from the 5-dimension sub-scores was applied and ranges from 0.000 to 1.000; higher scores indicate better patient-reported health status.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 136 | 136
units on a scale | .118 (.194) | .089 (.210)

12. Secondary Outcome: Number of Participants With Primary Patency
Description: Defined as freedom from clinically-driven target lesion revascularization (TLR) and freedom from restenosis determined by duplex ultrasound or angiogram greater than or equal to 50% stenosis.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 123 | 128
Participants | 99 | 87

13. Secondary Outcome: Number of Participants With Major Adverse Events (MAEs)
Description: as for outcome 2
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 143 | 140
Participants | 0 | 2

14. Secondary Outcome: Number of Participants With Clinically-driven Target Lesion Revascularization (TLR)
Description: as for outcome 6
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 144 | 141
Participants | 6 | 2

15. Secondary Outcome: Clinical Success ABI
Description: Defined as ankle-brachial index ABI reported at 12 months as change from baseline. The ABI is the ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery. Ideally, this ratio should be 1.0, but is often less in a subject with peripheral arterial disease.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 117 | 117
units on a scale | .19 (.20) | .23 (.24)

16. Secondary Outcome: Clinical Success Rutherford Category
Description: Defined as Rutherford Category reported at 12 months as change from baseline. Clinical scale identifying three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss. 0 is asymptomatic and 6 is ulcers/gangrene.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 134 | 130
units on a scale | -2.22 (1.08) | -2.32 (1.04)

17. Secondary Outcome: Clinical Success Quality of Life
Description: Defined by Quality of Life assessed by EQ5D questionnaire reported at 12 months as change from baseline. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The overall summary index (from Shaw et. al.) computed from the 5-dimension sub-scores was applied and ranges from 0.000 to 1.000; higher scores indicate better patient-reported health status.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 131 | 126
units on a scale | .090 (.202) | .074 (.208)

18. Secondary Outcome: Number of Participants With Primary Patency
Description: as for outcome 12
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 115 | 118
Participants | 81 | 63

19. Secondary Outcome: Number of Participants With Major Adverse Events (MAEs)
Description: as for outcome 2
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 119 | 120
Participants | 0 | 2

20. Secondary Outcome: Number of Participants With Clinically-driven Target Lesion Revascularization (TLR)
Description: as for outcome 6
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 125 | 122
Participants | 11 | 11

21. Secondary Outcome: Clinical Success ABI
Description: Defined as ankle-brachial index ABI reported at 24 months as change from baseline. The ABI is the ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery. Ideally, this ratio should be 1.0, but is often less in a subject with peripheral arterial disease.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 100 | 95
units on a scale | .20 (.21) | .21 (.26)

22. Secondary Outcome: Clinical Success Rutherford Category
Description: Defined as Rutherford Category reported at 24 months as change from baseline. Clinical scale identifying three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss. 0 is asymptomatic and 6 is ulcers/gangrene.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 107 | 111
units on a scale | -2.15 (1.14) | -2.12 (1.29)

23. Secondary Outcome: Clinical Success Quality of Life
Description: Defined by Quality of Life assessed by EQ5D questionnaire reported at 24 months as change from baseline. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The overall summary index (from Shaw et. al.) computed from the 5-dimension sub-scores was applied and ranges from 0.000 to 1.000; higher scores indicate better patient-reported health status.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
Number analyzed (Participants) | 108 | 108
units on a scale | .080 (.204) | .089 (.216)

ADVERSE EVENTS:
Time Frame: Follow-up data was collected through 24 months.
Arm/Group | Lithoplasty System Followed by DCB | Medtronic IN.PACT (DCB)
All-Cause Mortality (participants affected / at risk) | 17/153 | 12/153
Serious Adverse Events (participants affected / at risk) | 87/153 | 91/153
Other Adverse Events (participants affected / at risk) | 134/153 | 135/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lithoplasty System Followed by DCB (N=153) | Medtronic IN.PACT (DCB) (N=153)
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Empyema (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 2
Intervertebral discitis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 10
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 2
Septic shock (Infections and infestations) | 2 | 1
Staphylococcal infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Wound abscess (Infections and infestations) | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphocele (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 2 | 0
Lumbar spinal stenosis (Nervous system disorders) | 0 | 2
Peroneal nerve injury (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Sleep apnoea syndrome (Nervous system disorders) | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 2
Vertebral lateral recess stenosis (Nervous system disorders) | 1 | 0
Blepherochalasis (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 4
Glaucoma (Eye disorders) | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 5 | 4
Angina pectoris (Cardiac disorders) | 1 | 3
Angina unstable (Cardiac disorders) | 4 | 2
Aortic valve stenosis (Cardiac disorders) | 2 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 4
Cardiac failure chronic (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 4
Cardiogenic shock (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 7 | 6
Endocarditis (Cardiac disorders) | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 2
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Arterial bypass occlusion (Vascular disorders) | 1 | 0
Brain stem stroke (Vascular disorders) | 0 | 1
Carotid artery disease (Vascular disorders) | 1 | 0
Carotid artery stenosis (Vascular disorders) | 1 | 2
Cerebral infarction (Vascular disorders) | 0 | 2
Cerebrovascular accident (Vascular disorders) | 2 | 0
Coronary artery occlusion (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Iliac artery restenosis (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 1
Intermittent claudication (Vascular disorders) | 7 | 6
Intraventricular haemorrhage (Vascular disorders) | 0 | 1
Ischaemic stroke (Vascular disorders) | 1 | 2
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Penetrating aortic ulcer (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 6 | 4
Peripheral arterial reocclusion (Vascular disorders) | 4 | 2
Peripheral artery dissection (Vascular disorders) | 1 | 4
Peripheral artery occlusion (Vascular disorders) | 6 | 4
Peripheral artery restenosis (Vascular disorders) | 9 | 4
Peripheral artery stenosis (Vascular disorders) | 6 | 3
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1
Presyncope (Vascular disorders) | 0 | 2
Pulmonary embolism (Vascular disorders) | 0 | 1
Skin ulcer (Vascular disorders) | 2 | 3
Syncope (Vascular disorders) | 2 | 1
Transient ischaemic attack (Vascular disorders) | 1 | 0
Vascular graft occlusion (Vascular disorders) | 1 | 0
Vascular stent stenosis (Vascular disorders) | 3 | 1
Vascular stent thrombosis (Vascular disorders) | 0 | 1
Vertebrobasilar stroke (Vascular disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Helicobacter gastritis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 1
Phimosis (Reproductive system and breast disorders) | 1 | 0
Scrotal haematoma (Reproductive system and breast disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 3
Death (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Ureteroscopy (Investigations) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Atheroembolism (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Elastic vessel recoil complication (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Implant site infection (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 2
Aortic aneurysm repair (Surgical and medical procedures) | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Device breakage (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lithoplasty System Followed by DCB (N=153) | Medtronic IN.PACT (DCB) (N=153)
Pneumonia (Infections and infestations) | 6 | 12
Intermittent claudication (Vascular disorders) | 15 | 17
Peripheral arterial occlusive disease (Vascular disorders) | 36 | 26
Peripheral artery dissection (Vascular disorders) | 31 | 32
Peripheral artery occlusion (Vascular disorders) | 11 | 6
Peripheral artery restenosis (Vascular disorders) | 15 | 13
Peripheral artery stenosis (Vascular disorders) | 19 | 16
Coronary artery disease (Cardiac disorders) | 8 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 9
Atrial fibrillation (Cardiac disorders) | 8 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT02923193/Prot_SAP_000.pdf